CLINICAL TRIAL: NCT02242058
Title: Quantitative Sensory Testing and Pupillometry in Sickle Cell Disease Patients.
Brief Title: QST-Pupillometry in Sickle Cell Disease Patients
Acronym: QST
Status: Completed | Type: Observational
Sponsor: Julia Finkel (Other)
Responsible Party: Sponsor-Investigator, Julia Finkel, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: QST-Pupillo3614
Record Dates: First submitted 2013-09-13; First posted 2014-09-16 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: SCD With Severe Phenotype (HbSS, HbSβ0 Thalassemia, HbSOARab)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of blood samples at baseline to be stored in the Pain Neurobiology laboratory for future biochemical studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- High frequency pain group: 39 pediatric or adult patients with high pain frequency (greater than or equal to 3 ER visits and/or hospitalizations for pain per year over the last two years)
  Interventions: Other: Quantitative sensory testing
- Low Pain Frequency group: 39 pediatric or adult patients with low pain frequency (less than or equal to 1 severe pain episode for the last two years)
  Interventions: Other: Quantitative sensory testing
- Healthy control group: 39 pediatric or adult relatives of sickle cell disease patients, who do not have the sickle cell trait of SCD.
  Interventions: Other: Quantitative sensory testing
- Pain Crisis group: 30 patients with sickle cell disease with severe phenotype (HbSS, HbSβ0 thalassemia, HbSOArab)
  Interventions: Other: Quantitative sensory testing
- Pain Service group: 10 patients without sickle cell disease admitted to the pain service.
  Interventions: Other: Quantitative sensory testing

INTERVENTIONS:
Other: Quantitative sensory testing

SUMMARY:
There has been little progress for effective treatment of pain in sickle cell disease (SCD) patients. Many organizations have recognized that understanding the causes and reducing the burden of pain in SCD is critical in order to improve the quality of life in SCD patients. As patients with SCD face the challenge of living with both acute and chronic pain which is often improperly treated, our translational and interdisciplinary project aims to identify objective measures of pain sensitivity and its biochemical and genetic correlates. We hypothesize that SCD patients will have decreased tolerance to thermal and electrical stimuli.

ELIGIBILITY:
Inclusion Criteria:

* SCD with severe phenotype (HbSS, HbSbeta0 thalassemia, HbSOArab)
* Relatives of SCD patients who do not have sickle cell trait or SCD; healthy controls

Exclusion Criteria:

* Completed overt clinical stroke or transient ischemic attack;
* Known severe vasculopathy or Moyamoya disease on brain MRA (Magnetic Resonance Angiography).
* history of having consumed alcohol within the last 12 hours prior to testing.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: SCD patients referred to the Pain Medicine clinic, either outpatient or inpatient.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-08; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Measuring thermal responsiveness (perception and tolerance) in the outpatient groups. | change between baseline and at 90day follow-up
  Using a TSA (thermal sensory analyzer), the patients hot and cold perception and tolerance will be measured in the outpatient groups (high-pain and low-pain frequency and controls).
Measuring thermal responsiveness (perception and tolerance) in the inpatient groups. | change over 8 consecutive days
  Using a TSA thermal sensory analyzer, the patients hot and cold perception and tolerance will be measured in the inpatient groups (pain crisis and pain service).
Measure mechanical responsiveness in outpatient groups. | change between baseline and 90 day follow-up
  Using the Wagner PPIX 50 Pressure device, patient's tolerance to pressure is assessed in the outpatient groups (high-pain and low-pain frequency and controls).
Measure mechanical responsiveness in inpatient groups. | change over 8 consecutive days
  Using the Wagner PPIX 50 Pressure device, patient's tolerance to pressure is assessed in the inpatient groups (pain crisis and pain service).
Measuring the pupil responsiveness in outpatient groups. | change between baseline and 90 day follow-up
  Using the Pupillometer device, pupil responses are assessed in the outpatient groups (high-pain and low-pain frequency and controls).
Measuring the pupil responsiveness in inpatient groups. | change over 8 consecutive days
  Using the Pupillometer device, pupil responses are assessed in the inpatient groups (pain service and pain crisis).
Measuring electrical sensitivity in outpatient groups. | change between baseline and at 90day follow-up
  Using the Neurometer device, to assess electrical sensory perception and tolerance in the outpatient groups (high-pain and low-pain frequency and control).
Measuring electrical sensitivity in inpatient groups. | change over 8 consecutive days
  Using the Neurometer device, to assess electrical sensory perception and tolerance in the outpatient groups (pain service and pain crisis).

CONTACTS AND LOCATIONS:
Overall Officials: Julia Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Health System, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia